CLINICAL TRIAL: NCT02867644
Title: Randomized Trial Comparing the Contribution of Conversational Hypnosis Versus Standard Care on Patient Anxiety During a Preoperative Breast Tracking
Brief Title: Conversational Hypnosis in Women Undergoing Imaging for Breast Cancer
Acronym: HYCOREMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Results not achievable after interim analysis conclusions and recruting difficulty
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-A00232-49
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
Keywords: conversational hypnosis; imaging; care; breast neoplasia; anxiety; pain
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care (Active Comparator)
  Interventions: Other: standard care
- standard care+conversational hypnosis (Experimental)
  Interventions: Other: standard care + conversational hypnosis

INTERVENTIONS:
Other: standard care — Patients coming for preoperative breast assessment will have standard care.
  Arms: standard care
Other: standard care + conversational hypnosis — Patients coming for preoperative breast assessment will have standard care with conversational hypnosis
  Arms: standard care+conversational hypnosis

SUMMARY:
The hypothesis is to assess the contribution of conversational hypnosis on anxiety of patients who undergoing for a preoperative breast tracking and improve their care

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patient undergoing for a preoperative breast assessment
* Patient must be affiliated to a social security system
* Ability to provide an informed written consent form

Exclusion Criteria:

* Patients diagnosed with major hearing loss
* Patients with schizophrenia
* Patients do not understand the French language
* Pregnant or breast feeding females
* Refusal of the patient to participate in the study
* Persons deprived of liberty or under supervision

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Compare anxiety of patients undergoing for a preoperative breast marking under ultrasound according two different procedures (standard care versus standard care with conversational hypnosis) | Day 1
  The anxiety level will be assessed in each group by a visual analog scale from 0 to 10.

SECONDARY OUTCOMES:
Compare the pain felt by patients during a preoperative breast marking under ultrasound according two different procedures (standard care versus standard care with conversational hypnosis) | Day 1
  The pain level will be assessed in each group by a visual analog scale from 0 to 10.
Compare the manipulator's satisfaction during a preoperative breast marking under ultrasound according two different procedures (standard care versus standard care with conversational hypnosis) | Day 1
  The manipulator's satisfaction will be assessed in each group by a numeric scale from 0 to 10.
Evaluate the receptivity of women to conversational hypnosis | Day 1
  assessment realisation time flet by patient
Assess the impact of conversational hypnosis on completion of the examination | Day 1
  The assessment will be evaluated in each group by the radiologist according to a visual analog scale from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: HENROT Philippe, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (7):
- France (7):
  - CH Bastia, Bastia
  - Chu Bordeaux-Pellegrin, Bordeaux
  - CHRU de Brest, Brest
  - Centre Léon Bérard, Lyon
  - APHM La Timone, Marseille
  - Centre Paul Strauss, Strasbourg
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lemoine L, Adam V, Galus X, Siles P, Coulon A, Grenier-Desforges J, Orabona J, Kergastel I, Wagner P, Salleron J, Tosti P, Huin-Schohn C, Merlin JL, Etienne R, Henrot P. Conversational hypnosis versus standard of care to reduce anxiety in patients undergoing marker placement under radiographic control prior to breast cancer surgery: A randomized, multicenter trial. Front Psychol. 2022 Nov 22;13:971232. doi: 10.3389/fpsyg.2022.971232. eCollection 2022. PMID 36483698